CLINICAL TRIAL: NCT05239663
Title: The Effects of Ganglioside-Monosialic Acid in Post-chemotherapy Cognitive Impairment in Patients With Early Operable Breast Cancer: A Randomized Trial
Brief Title: GM1 Prophylaxis for Post-chemotherapy Cognitive Impairment in Patients With Early Operable Breast Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty accruing subjects the study accrual was closed
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Zhong-yu Yuan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SYSUCC-016
Record Dates: First submitted 2022-02-07; First posted 2022-02-15 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Chemotherapy-Related Cognitive Impairment; Breast Cancer
Keywords: Ganglioside-Monosialic Acid, post-chemotherapy cognitive impairment, breast cancer
MeSH Terms: conditions — Chemotherapy-Related Cognitive Impairment; Breast Neoplasms | interventions — Neuroprotective Agents; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): standard (neo)adjuvant chemotherapy plus Ganglioside-Monosialic Acid 100mg+250ml normal saline (NS)
  Interventions: Drug: Ganglioside-Monosialic Acid
- Control group (Other): standard (neo)adjuvant chemotherapy plus 250ml normal saline (NS)
  Interventions: Drug: 250ml normal saline (NS)

INTERVENTIONS:
Drug: Ganglioside-Monosialic Acid — Standard (neo)adjuvant chemotherapy (Taxanes combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by taxanes) plus Ganglioside-Monosialic Acid 100mg+250ml normal saline (NS)
  Other Names: neuroprotective agents
  Arms: experimental group
Drug: 250ml normal saline (NS) — Standard (neo)adjuvant chemotherapy (Taxanes combined with cyclophosphamide or doxorubicin combined with cyclophosphamide followed by taxanes) plus 250ml normal saline (NS)
  Other Names: placebo
  Arms: Control group

SUMMARY:
The purpose of this study is to evaluate the prophylactic effects of Ganglioside-Monosialic Acid in post-chemotherapy cognitive impairment in patients with early operable breast cancer.

DETAILED DESCRIPTION:
This is a multicenter, prospective, randomized, single-blind, phase III clinical trial. The primary endpoint is the changes of cognitive function from baseline to 4 weeks after the completion of adjuvant chemotherapy in the experimental group and the control group, which were evaluated by HVLT-R scale. This study is designed to recruit up to 306 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Have provided written and signed informed consent;
2. Histologically confirmed invasive ductal carcinoma;
3. Planned to received (neo)/adjuvant chemotherapy;
4. Eastern Cooperative Oncology Group (ECOG) score of 0 to 1;
5. Can cope with HVLT-RDR and ADAS-Cog evaluation;
6. No prior therapy could induce neurological damage,within 4 weeks
7. Normal blood routine, liver and kidney functions within 1 week before enrollment in this study;
8. Women of childbearing age have a negative serum or urinary pregnancy tests prior to enrollment in this study; Pre-menopause women are contracepted with medically acceptable methods during the study period.
9. Compliance with the study protocol.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) score ≥ 2;
2. Hypersensitivity to experiment agents or components;
3. Women with pregnancy or breast feeding;
4. A clear past history of neurological or psychiatric disorders, including epilepsy or dementia;
5. Abnormal baseline impairment of cognitive impairment;
6. Poor compliance, unwillingness or inability to follow protocol to continue the study;
7. Any circumstances in which the investigator deemed the subject unsuitable for enrollment in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-02-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
HVLT R-DR | 4 weeks after the completion of adjuvant chemotherapy
  The change of score for Hopkins verbal learning test -revised,delayed recall,from baseline to 4 weeks after the completion of adjuvant chemotherapy.

SECONDARY OUTCOMES:
HVLT R-DR | 36 weeks after the completion of adjuvant chemotherapy
  The change of score for Hopkins verbal learning test -revised,delayed recall,from baseline to 12 weeks，24 weeks and 36 weeks after the completion of adjuvant chemotherapy.
ADAS-Cog | 36 weeks after the completion of adjuvant chemotherapy
  The change of score for Alzheimer's Disease Assessment Scale-Cognitive,from baseline to 12 weeks，24 weeks and 36 weeks after the completion of adjuvant chemotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China